CLINICAL TRIAL: NCT06746571
Title: Role of Cbc Indices in Acute Lymphoblastic Leukemia Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Omnia Aly Mohamed, resident-clinical pathology sohag university hospital, Sohag University
Allocation: Not Applicable | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: soh-MED--24-12-09ms
Record Dates: First submitted 2024-12-18; First posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Blood Cell Count

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: complete blood count — measure cbc and blood ratios to compare their values with respone of patients to treatment

SUMMARY:
Role of cbc indices in acute lymphoblastic leukemia patients to explore the prognostic role of them in prediction the response to induction chemotherapy

DETAILED DESCRIPTION:
Role of neutrophil to lymph ratio , lymphocyte to monocyte ratio and platelet to lymphocyte in acute lymphoblastic leukemia adults and pediatric patients to explore the prognostic role of them in prediction the response to induction chemotherapy

ELIGIBILITY:
Inclusion Criteria:

* patients newly diagnosed ALL

Exclusion Criteria:

* others malignanices
* ALL on therapy

Ages: 5 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
neutrophil to lymphocyte ratio | 1 year
  count of neutophils comparing lymphocytees

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jiang Z, Dong Z, Wang L, Jiang W. Method for Diagnosis of Acute Lymphoblastic Leukemia Based on ViT-CNN Ensemble Model. Comput Intell Neurosci. 2021 Aug 21;2021:7529893. doi: 10.1155/2021/7529893. eCollection 2021. PMID 34471407
- [Background] Gavralidis A, Brunner AM. Novel Therapies in the Treatment of Adult Acute Lymphoblastic Leukemia. Curr Hematol Malig Rep. 2020 Aug;15(4):294-304. doi: 10.1007/s11899-020-00591-4. PMID 32445026
- [Background] Haider RZ, Ujjan IU, Khan NA, Urrechaga E, Shamsi TS. Beyond the In-Practice CBC: The Research CBC Parameters-Driven Machine Learning Predictive Modeling for Early Differentiation among Leukemias. Diagnostics (Basel). 2022 Jan 7;12(1):138. doi: 10.3390/diagnostics12010138. PMID 35054304
- [Background] Stefaniuk P, Szymczyk A, Podhorecka M. The Neutrophil to Lymphocyte and Lymphocyte to Monocyte Ratios as New Prognostic Factors in Hematological Malignancies - A Narrative Review. Cancer Manag Res. 2020 Apr 29;12:2961-2977. doi: 10.2147/CMAR.S245928. eCollection 2020. PMID 32425606